CLINICAL TRIAL: NCT01424280
Title: A Phase 1, Randomized, Placebo Controlled, Crossover Study to Evaluate the Efficacy of GSK1440115 After a Single Oral Dose in Patients With Asthma
Brief Title: Single Dose Study of GSK1440115 in Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UR2115642
Record Dates: First submitted 2011-08-01; First posted 2011-08-26 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — 4'-(1-(((6,7-dichloro-3- oxo-2,3-dihydro-4H-1,4-benzoxazin-4-yl)acetyl)(methyl)amino)-2-(4-morpholinyl)ethyl)-4-biphenylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Experimental)
  Interventions: Drug: 1440115
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1440115 — Single dose of either 750 mg or 500 mg administered as 250 mg tablets.
  Arms: Active drug
Drug: Placebo — Single dose of matching placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess bronchodilator effect after single dose administration of GSK1440115 in a population of mild to moderate asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Male or female between 18 and 65 years of age, inclusive, at the time of signing informed consent.
3. Male patients with a female partner of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of study drug until three months after the last dose of study drug.
4. A female patient is eligible to participate if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods defined in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least two to four weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   2. Child-bearing potential, has a negative serum pregnancy test during the Screening Period, and agrees to use adequate contraception from Screening until four weeks after the last dose of study drug.
5. BMI within the range of 19-32 kg/m2 (inclusive).
6. Documented history of bronchial asthma that is British Thoracic Society guideline step 1-3, diagnosed at least 3 months prior to the Screening visit.

   a. Patient should be on a fixed regimen for at least 4 weeks prior to Screening. The following asthma medications are permitted: i. Inhaled corticosteroid (ICS) per day use: <=800mcg of Beclomethasone Dipropionate or budesonide, 320mcg ciclesonide or 500mcg of Fluticasone propionate - or equivalent doses.

   ii. Intermittent short-acting inhaled beta-2 agonist therapy (SABA). A minimum of 8 hours washout from SABA is required prior to Screening or study methacholine challenge tests or FEV1 assessments.

   iii. Long-acting inhaled beta-2 agonist (LABA) therapy is not permitted during the study. If deemed appropriate by the investigator, patients usually managed with LABA can be switched to SABA in order to comply with requirements for washout. A minimum of 24 hour washout after last dose of LABA is required prior to Screening methacholine challenge tests or FEV1 assessments.

   iv. Therapy with montelukast is allowed provided that administration is separated by at least 12 hours from study drug dosing (see Section 9).
7. Best FEV1 of >70% predicted normal value during Screening.
8. Hyper-responsive to methacholine such that a baseline methacholine PC20 is <= 4 mg/mL.
9. Increase in PC20 of at least 2 dilutions compared to baseline in the presence of inhaled beta-agonist in response to a methacholine challenge.
10. Patients who are currently non-smokers or who have not used any inhaled tobacco products in the previous 6 months prior to first dose of study drug.
11. Average QTcF < 450 msec; or QTc < 480 msec in patients with Bundle Branch Block.
12. AST and ALT < 2xULN; alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening.
2. A positive test for HIV antibody.
3. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. A positive pre-study drug/alcohol screen.
5. History of regular alcohol consumption within 6 months of the study defined as:

   History of regular alcohol intake (average weekly intake of > 21 units males or >14 units females - One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.
6. History of chronic medical disease that in the investigators opinion may affect the outcome of the study - including interpretation of safety data. This may include, but is not limited to, malignancy, cardiovascular, hepatic, renal, hematological, neurological, thyroid disease, endocrine disease, or, other pulmonary diseases. Examples of specific exclusions include:

   * History of heart attack or stroke within past 3 months.
   * Presence of known aortic aneurysm.
   * Epilepsy.
   * COPD, pulmonary fibrosis, or bronchiectasis
   * Peptic ulcer disease.
   * Urinary tract obstruction.
7. Clinically significant laboratory abnormalities at Screening.
8. History of uncontrolled hypertension or persistent SBP>140 mmHg or DBP >90mmHg at Screening.
9. History of life-threatening asthma (asthma episode requiring intubation and/or associated with hypercapnea, respiratory arrest or hypoxic seizure) OR the following:

   * Respiratory tract infection and/or asthma exacerbation within 4 weeks prior to the first dose of study drug.
   * Asthma exacerbation requiring hospitalization within 3 months prior to Screening.
   * Administration of systemic steroids within 4 weeks of Screening.
10. Intake of an investigational product within either 30 days or 5 half lives (whichever is longer) prior to first dose of study drug.
11. History of sensitivity to any of the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
12. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
13. Lactating females.
14. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to Screening.
15. Current use of a prohibited medication or requires use of a prohibited medication during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Methacholine PC20 | 7 hours post dose

SECONDARY OUTCOMES:
Change from baseline in FEV1 | 1, 2, 3, 4, 5, 6, and 7 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, New South Wales, Australia